CLINICAL TRIAL: NCT05608707
Title: Innovative PlAnt Protein Fibre and Physical Activity Solutions to Address Poor AppEtite and PrevenT UndernutrITion in OldEr Adults (APPETITE)
Brief Title: APPETITE: Plant Protein and Exercise Solutions for the Prevention of Undernutrition in Older Adults.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: LS-21-96-Roche; JPI-ERA-HDHL PREVNUT-2020-1 (Other Grant/Funding Number: Health Research Board (HRB))
Record Dates: First submitted 2022-10-10; First posted 2022-11-08 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Appetite Loss; Physical Inactivity; Undernutrition; Anorexia of Aging; Aging; Ageing Well
Keywords: appetite; energy intake; nutrition; older adults; Physical activty
MeSH Terms: conditions — Anorexia; Sedentary Behavior; Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial, a two-by-two factorial design will define the individual and combined impact of two intervention conditions over 12 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Personalised diet plus physical activity intervention (Experimental): A personalised diet intervention involving the incorporation of the developed plant-based protein and fibre product.
  Participants will also undertake 2 weekly group exercise sessions incorporating strength and balance exercises, along with home-based exercise
  Interventions: Behavioral: Physical activity intervention; Dietary Supplement: Personalised nutrition intervention
- Usual diet plus physical activity (Experimental): Participants will consume their usual diet and undertake 2 weekly group exercise sessions incorporating strength and balance exercises, along with home-based exercise
  Interventions: Behavioral: Physical activity intervention
- Personalised diet plus usual physical activity (Experimental): A personalised diet intervention involving the incorporation of the developed plant-based protein and fibre product.
  Interventions: Dietary Supplement: Personalised nutrition intervention
- Control (usual diet and physical activity) (No Intervention): This arm will not be given any nutritional or physical activity support. They will be instructed to carry on with their usual activities.

INTERVENTIONS:
Behavioral: Physical activity intervention — The 12 week intervention will involve 2 weekly group exercise sessions incorporating strength and balance exercises, along with home-based exercise focused on increasing time spent walking.
  Other Names: Structured exercise program
  Arms: Personalised diet plus physical activity intervention; Usual diet plus physical activity
Dietary Supplement: Personalised nutrition intervention — Two Plant-based Protein and Fibre (PPF) product products have been selected from six initially developed, with best amino acid blend, taste, and bioavailability. Participants will be provided with the PPFs to consume daily as part of a personalised diet over 12 weeks.
  Other Names: Plant-based protein and fibre intervention
  Arms: Personalised diet plus physical activity intervention; Personalised diet plus usual physical activity

SUMMARY:
The APPETITE Trial aims to investigate the efficacy of innovative plant protein fibre (PPF) products (developed in a previous workpackage) as part of a personalised diet with/out physical activity on appetite and incidence of undernutrition in older persons from three European countries at high risk of undernutrition.

DETAILED DESCRIPTION:
It is normal that dietary intake decreases as we age due to reduced activity and muscle mass. However, appetite is a key determinant of dietary intake, and poor appetite can result in undernutrition. In many instances, older adults do not recognise their appetite has decreased significantly as the decline is slow and progressive. Protein and fibre are often poorly consumed in the diets of older adults with decreased appetite, but essential for health and well-being. Interventions designed to increase appetite, or increase dietary intake despite a reduced appetite, should therefore be key to preventing undernutrition (i.e. protein-energy malnutrition as well as nutrient deficiencies). However, treatment strategies for poor appetite are not well-established.

In this multi-centre randomised controlled trial conducted in Ireland, Germany, and Italy, a two-by-two factorial design will define the individual and combined impact of two intervention conditions over 12 weeks: 1) personalised diet with focus on plant-based protein plus fibre; and 2) physical activity.

At each centre, 60 older adults (180 in total) will be randomly allocated to one of the following four groups over a 12 week period: 1) personalised diet plus physical activity program (PD + PA), 2) usual diet plus physical activity (PA), 3) personalised diet and no PA (PD), and 4) control (usual diet, no PA).

Using identical procedures, two testing visits will be completed before and after the 12 intervention or control period.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling,
* Age 65+ years,
* BMI 19.5-30.4kg/m2,
* Inactive (<150 minutes of moderate to vigorous physical activity per week and no regular resistance training),
* Have proof of Covid-19 vaccination

Exclusion Criteria:

* Major cognitive impairment (MMSE ≤24),
* Uncontrolled Clinical depression (CES-D >16),
* Medical condition or current medication known to impact appetite or energy intake,
* Other medical condition that may impact ability to participate in study or study outcomes,
* Heavy smoker (>10/day),
* Plans to relocate out of the study area within the next 6 months,
* Inability to come to study centre/PA program location,
* Currently participating in another intervention study,
* Inability to participate in physical activity,
* Unable to walk across a room,
* Allergic to or unwilling to consume any of the study test foods,
* Loss of taste or smell associated with COVID-19,
* Unwilling to be randomised to any intervention group.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Ad libitum energy intake (kcal) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in energy intake assessed at an an ad libitum lunch test meal
Changes in subjective appetite sensations | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in appetite to be assessed by Visual Analogue Scale (VAS) during a test meal challenge. The VAS is a validated tool for assessing subjective sensations such as hunger, fullness and desire to eat. On each 100-mm line, an appetite (hunger, fullness, desire to eat) sensation was paired with the opposing sensation (for example, 'hungry' and 'not hungry').

SECONDARY OUTCOMES:
7-day physical activity score as assessed by ActivPAL v4.0 | To be assessed at baseline, prior to commencing the intervention, and during week 12 of the intervention or control period
  12-week change in physical activity score will be assessed using 7-day accelerometery data. This is a validated device that is installed onto an individuals thigh for continuous readings. The data generated describes the amount of time spent engaging in physical activities and sedentary activities, and gives an output score in MET.h (Metabolic EquivalenT hour). This is a measure of energy usage over and above what is required at rest, where 1MET is equivalent to oxygen uptake of 3.5ml/kg body weight/minute
Resting Energy Expenditure (REE) (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in resting energy expenditure will be assessed using indirect calorimetry
Handgrip strength | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in handgrip strength will be assessed using a Jamar hydraulic hand dynamometer
Isometric knee extension strength | To be assessed at baseline and following a 12-week intervention or control period
  12-week changes in isometric leg strength will be assessed using a seated leg extension dynamometer
Cardiorespiratory fitness | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in cardiorespiratory fitness will be assessed using the 400-meter walk test
Physical performance | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in physical function will be assessed using the Short Physical Activity Battery (SPPB)
Participants subjective rating of perceived Quality of Life as assessed by the EQ-5D-5L | To be assessed at baseline and following a 12-week intervention or control period
  12-week changes in perceived quality of life will be assessed using the EuroQol (European Quality Of Life) questionnaire (EQ-5D-5L). This consists of self-assessed rating of health under 5 dimensions (Mobility, Self-Care, Usual Activity, Pain/Discomfort, Anxiety/Depression), and perceived overall health on a magnitude scale (0-100) anchored with opposing statements (0= the worst health you can imagine; 100= the best health you can imagine).
Body composition (fat mass, fat free mass) by air displacement phlethysmography (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in body composition will be assessed using air displacement plethysmography (Bodpod).
Cognitive Dietary Restraint | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in dietary restraint will be assessed using the Cognitive Dietary Restraint (CDR) subscale of the Three Factor Eating Questionnaire (TFEQ). The questionnaire consists of a subscale of 6 questions relating to cognitive dietary restraint from the orignal 50 item questionnaire. The questions are a mix of 'true/false', and likert scale type answers.
Dietary Record (energy, protein and fibre intake) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in energy, protein and fibre intake assessed using a three-day non-weighed dietary record
Appetite hormones (Ghrelin, GLP-1, & PYY) (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in appetite-related gut hormone response to a fixed meal. Assessed in circulating peripheral bloods at fasting, and at regular intervals postprandially (minute 30, 60, 90, 120, 150, & 180).
Gut metabolomic profiles and gut microbiome diversity | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in gut microbiota quality and diversity assessed by faecal matter and faecal water.
Blood hormone and metabolite profile | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in fasting peripheral blood profile (insulin, leptin, glucose, amino acid, fatty acid)
Body composition by Bioelectrical Impedance Analysis (BIA) | To be assessed at baseline and following a 12-week intervention or control period
  Body composition will be assessed by BIA across all sites at baseline and post intervention. BIA is a quick non-invasive method of measuring body composition. Bioelectrical impedance analysis (BIA) measures body composition based on the rate at which an electrical current travels through the body. Body fat (adipose tissue) causes greater resistance (impedance) than lean mass and slows the rate at which the current travels. The device provides an output of absolute (Kg) and percentage (% of total mass) of fat mass (FM) and fat-free mass (FFM).
Appetite by Simplified Nutritional Appetite Questionnaire (SNAQ) | To be assessed at baseline and following a 12-week intervention or control period
  The SNAQ questionnaire is used to assess an older adults usual appetite. The SNAQ is a self-administered questionnaires adapted from the Appetite, Hunger and Sensory Perception questionnaire (AHSP), an appetite assessment tool validated among community-dwelling older adults. It consists of 4 multiple choice statements, where an individual reads the beginning of the statement and is presented with 5 options that best describe their situation. Each question derives a score between 1 - 5 with lower scores indicating poorer appetite. The questionnaire scores between 4 - 20 with scores </= 14 indicating poor appetite.
Test meal palatability by Visual Analogue Scale (VAS) | To be assessed at baseline and following a 12-week intervention or control period
  Rating of the breakfast and lunch test meals by visual analogue scales (VAS). The VAS is a validated tool for assessing subjective sensory experience. On each 100-mm line, a question is asked relating to sensory aspects of the meal (E.g., How pleasant was the meal?). The subject will mark along the 100mm line where they feel their experience, in terms of the question, rests. On ether end of the 100mm line are opposing terms (E.g., "not at all", "extremely").
Body weight (kg) | To be assessed at baseline and following a 12-week intervention or control period
  Body weight will be measure using a calibrated scales, shoes and heavy clothing removes, and recorded in kilograms.
Standing height (cm) | To be assessed at baseline and following a 12-week intervention or control period
  Height will be measured in centimetres using a stadiometer. Participants will be measured barefoot and asked to take a full inhalation prior to stepping out from the device. Measurements are taken at the peak of the inhalation.
Calf circumference (cm) | To be assessed at baseline and following a 12-week intervention or control period
  Calf circumference is measures using a non-stretch tape measure at the widest part of the calf muscle and recorded in centimetres.
Perception and evaluation of the trial | End of trial (up to 18-weeks)
  Questionnaire specific to the project. This questionnaire will serve to provide feedback about participants experience while enrolled on the project. The questionnaire will include a series of Likert style questions and open-ended questions. The purpose is the provide feedback to the study team on what participants liked or disliked about the experience. This will serve to inform future management of studies.
Body composition by Dual-energy X-ray absorptiometry (DXA) (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  DXA will be performed on a sub-sample of participants enrolled on the APPETITE study. A DXA can involves a large scanning arm being passed over the body to measure compartments of the body structure. As the scanning arm is moved slowly over your body, a narrow beam of low-dose X-rays will be passed through the part of your body being examined. DXA is a quick and non-invasive scan that provides in-depth analysis of the main components of your body; fat, muscle and bone.
Motor Unit Signalling (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  by electromyography (EMG)
Motor Unit Number | To be assessed at baseline and following a 12-week intervention or control period
  from muscle biopsy
muscle signalling related to muscle plasticity, metabolism, denervation and muscle capillarization (sub-sample) | To be assessed at baseline and following a 12-week intervention or control period
  This refers to the analyses of muscle biopsies. Biopsies will be taken using MEDAX/BF14100-C0; Bio-Feather with coaxial 14 g 10 cm. The following parameters will then be measured in the sample using western blot with specific antibodies for total proteins or by their activated phosphorylated form: 1) markers of denervation (AChR ; agrin/MuSK/Lrp4, NCAM, Myog); 2) markers of protein turnover (atrogin1, MURF1, LC3, BNIP3, Akt-dependent mTOR and FoxO); 3) markers of mitochondrial dynamics (OPA1, DRP1) and; 4) markers of energy metabolism pathways (AMPK and PGC1alpha).
Innate immune training of macrophages | To be assessed at baseline and following a 12-week intervention or control period
  Trained immunity describes the long-term functional reprogramming of innate immune cells after exposure to a primary insult which leads to an augmented response upon stimulation with the same ligand after returning to a non-activated state. Will habitual ingestion of plant protein combined with PA results in increased ability of macrophages to undertake innate immune train in adults over the age of 65. Effects will be quantified by comparing the presence of TNF alpha in human monocytes at baseline and following a 12-week intervention.

OTHER OUTCOMES:
Physical Activity Scale for the Elderly (PASE) | To be assessed at baseline and following a 12-week intervention or control period
  Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older
Adherence and acceptability of the intervention | Throughout intervention
  Adherence to the intervention requirements will be assessed using compliance diaries. Participants will record in a diary, provided by the study team, each time they consume the study product and/or complete a physical activity session. They will also collect empty sachets and return them to the study team at the end of the intervention. Compliance is considered adequate if 10 of a possible 14 supplements per week are consumed, and/or attendance of >80% structured physcial activity sessions.
Self-efficacy in adhering to the intervention | At baseline
  This will take the form of a couple of questions during initial screening. The purpose of these questions is to assess whether the participant believes they can fulfil the intervention requirements if enrolled onto the study. The logic is to identify those who are unlikely to complete the study as a mechanism of reducing dropout rates. The questions will take the form of a Likert scale, and relate to the participants confidence, or lack thereof, to complete key requirements of the study.
Cognitive status by Mini Mental State Examination (MMSE) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in global cognition assessed by Mini Mental State Examination (MMSE). The MMSE is a commonly used tool to exam global cognition in both clinical and research setting. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score for the MMSE is 30 points, where scores <24 would be indicative of cognitive dysfunction.
Depressive symptoms assessed by Centre of Epidemiology Study - Depression (CES-D) | To be assessed at baseline and following a 12-week intervention or control period
  12-week change in depressive (Centre of Epidemiology Study - Depression) symptoms. The CES-D is a 20-item measure that rate how often over the past week an individual experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. A score equal to or greater than 16 is indicative of risk of clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Roche, Professor, Principal Investigator — UCD; Katy Horner, PhD, Principal Investigator — University College Dublin; Marjolein Visser, PhD, Principal Investigator — VU Amsterdam
Locations (3):
- FAU, Nuremberg, Germany
- School of Public Health, Physiotherapy and Sports Science, Dublin, Leinster, Ireland
- UNIPD, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horner KM, Mullen B, Quinn A, Scheufele P, Gola S, Gonnelli F, Bozzato M, Pratt J, Sala W, Mullin S, Kirwan L, Dardevet D, Guillet C, De Vito G, Visser M, Volkert D, Corish CA. Plant protein, fibre and physical activity solutions to address poor appetite and prevent undernutrition in older adults: study protocol for the APPETITE randomised controlled trial. Br J Nutr. 2024 Sep 28;132(6):823-834. doi: 10.1017/S0007114524002125. Epub 2024 Oct 10. PMID 39387205
- See also: Study specific website — https://www.jpi-appetite.com/
- See also: Study protocol paper — https://pmc.ncbi.nlm.nih.gov/articles/PMC11557289/